CLINICAL TRIAL: NCT07011563
Title: Prepping for The Talk: Helping Trusted Adults and Youth Talk About Sexual Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jack Rusley, Associate professor, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1554023; K23MH123335 (NIH)
Record Dates: First submitted 2025-06-05; First posted 2025-06-09 (Actual); Last update posted 2025-06-09 (Actual); Status verified 2025-06

CONDITIONS: HIV Prevention; Sexual Health
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Intervention
- Treatment as usual + (Active Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention — Youth: interventionist-facilitated 1:1 conversation with the youth via videoconference that includes a) brief sexual health assessment, b) individualized information about HIV risk reduction including PrEP, and c) use of motivational interviewing strategies to discuss barriers to PrEP.
  Parents: brief (~20-30 min) web-based, interactive learning module ("module") designed to provide information about sexual health communication (SHC) best practices, HIV prevention strategies (e.g., condoms, STI testing, PrEP), as well as build practical skills around SHC using evidence-based behavior change methods (e.g., building confidence, aligning values with actions).
  Arms: Intervention
Behavioral: Control — Youth: interventionist-facilitated 1:1 conversation with the youth via videoconference that includes a) brief sexual health assessment, and b) didactic information about condom use, STI testing (including HIV), and PrEP (but not motivational interviewing or individualized information on HIV risk reduction).
  Parent: brief written information on a digital platform (i.e., website) with advice about talking to youth about sexual health with web-links to resources about STI/HIV prevention and PrEP. This information will not be interactive or use behavior change methods.
  Arms: Treatment as usual +

SUMMARY:
The goal of this study is to help young people talk to trusted adults (including their parents, but also other adults) about sexual health more openly and honestly- including how to prevent sexually transmitted diseases like HIV - while also respecting a young person's right to privacy. If youth don't have a parent they can talk to about sexual health, we want to help them find a trusted adult to talk to. We also want to help youth take control of their own health by learning about different ways to protect their health.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-17
* Assigned male
* Oral OR anal sex with an assigned male
* Live in the United States
* English-speaking

Exclusion Criteria:

* None

Ages: 14 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Sexual health communication scale score - youth | 4 weeks
  We will administer the SHC scale to youth as a survey
Sexual health communication scale score - parent | 4 weeks
  We will administer the SHC scale to parent as a survey

SECONDARY OUTCOMES:
PrEP uptake | 4 weeks
  Self-reported initiation of PrEP by youth

CONTACTS AND LOCATIONS:
Overall Officials: Jack Rusley, MD, MHS, Principal Investigator — Brown University Health
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States